CLINICAL TRIAL: NCT00145860
Title: Do Patients With Colorectal Cancer Understand That Their Family is at Increased Risk?
Brief Title: Do Patients With Colorectal Cancer Understand That Their Family is at Risk?
Status: Terminated | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 11589A
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to assess whether patients with colorectal cancer understand that their first-degree relatives are at increased risk of getting the cancer themselves and therefore should be screened early. Among patients who do understand the risks to their family, we plan to determine who they identify as the source of their information and whether they have acted upon this information and advised family members to be screened. We hypothesize that many patients with colorectal cancer do not have a correct understanding of the risks to their first-degree relatives and the recommendations that they be screened early.

If this hypothesis is shown to be true, it can be used to direct improved and more diligent patient education. This, in turn, will hopefully increase the low screening rates among first-degree relatives, and, thereby, save lives in this high-risk population.

DETAILED DESCRIPTION:
1. The primary physician of patients with colorectal cancer will be contacted and asked permission to contact their patient to discuss his or her understanding of familial risk before patient is contacted.
2. A letter will be sent to all patients prior to being contacted, notifying them that all identifying information will be kept confidential and they may decline to participate at any time.
3. Patients will be called and asked a series of questions about their understanding of familial risk of colon cancer, the need for early screening and where they learned what they know. If the patient has lacking knowledge they will be educated.
4. Each patient will be sent informational brochures about colon cancer after the phone survey.
5. Six months later, the patients will be contacted again and asked a series of questions about their understanding of familial risk of colon cancer and the need for early screening to access how much impact the informational brochures had on their knowledge of cancer risk. Patients will be asked one additional demographic question about the highest level of education that they have completed.

ELIGIBILITY:
Inclusion Criteria:

Patients who were diagnosed with CRC and received first treatment here or elsewhere and patients who were diagnosed elsewhere and received their first treatment here. All are currently followed here and still alive.

Exclusion Criteria:

Patients in the registry who are not followed here, patients with Familial Adenomatous Polyposis, patients with Hereditary Non-Polyposis Colorectal Cancer, and patients with no siblings or children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2002-04; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: David Rubin, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States